CLINICAL TRIAL: NCT04034888
Title: Home Exercise Program for Homebound Older Adults
Acronym: HEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Alyssa Stookey, Research Health Scientist (GRECC), Research Associate (SOM), University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMaryland
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Exercise Program (HEX) (Experimental): Customized home exercise program
  Interventions: Behavioral: HEX

INTERVENTIONS:
Behavioral: HEX — HEX is a customized exercise program with components including: 1) controlled flexibility movements; 2) progressive ADL training focusing on bed mobility, bed to chair transfers, and indoor walking; 3) task-specific seated resistance training to improve ability to get out of bed and; 4) and balance exercises. Participants will be expected to perform their HEX program at least 2 times/week in their home and all individualized exercise sessions will be supervised by an Exercise Physiologist. Each exercise has four levels of difficulty, which will be progressed as tolerated throughout the 12-weeks. Seated resistance exercises were designed to target all the major muscle groups and will include the following: arm curls, shoulder raises (lateral/front), overhead arm raise, wrist curls, leg extensions, hip flexion, hip ab/adduction, sit-to-stands, torso rotation, and marching.

SUMMARY:
Exercise can be beneficial for older adults by promoting health, delaying or reversing functional decline, reducing chronic disease risk, decreasing falls, increasing strength and stamina, improving ability to perform activities of daily living (ADL), and improving overall quality of life (QOL). Developing and implementing exercise programs for homebound older adults for whom traveling to routine clinic-based appointments may not be feasible or safe becomes critical. Homebound, older adults are at increased risk for recurrent hospitalization, use of emergency care, nursing home placement, and death. Indeed, one study shows patients had significantly higher risk of being admitted into a hospital or nursing home, higher mortality, and higher health care expenditures compared to those in a comparison group. The purpose of this pilot is to develop and implement a pragmatic and feasible intervention to improve physical functioning in older homebound adults with chronic mobility disability. Unfortunately, little is known about the feasibility and utility of pragmatic home-based exercise rehabilitation in older adults with severe mobility limitations.

The investigators propose to develop and implement an intervention targeting functional limitations in this population with mobility disability. Our overall goals are to maintain and restore physical functioning and QOL for older, homebound adults. This research carries direct benefits for these patients as even modest improvements in disabled older adults may translate into significantly better QOL, reduce disability, minimize or reverse gradual declines related to serious chronic disease, resort functional independence, and increase community living capacity. Thus, the specified objectives of finalizing and implementing a sustainable home-based exercise program have practical implications for disabled older adults. Were homebound patients even slightly higher in terms of functional capacity, it could provide a partial degree of functional independence, impacting QOL for both patients and caregivers.

DETAILED DESCRIPTION:
The purpose of this study is to develop and implement a pragmatic and feasible intervention to improve physical functioning in older homebound adults with chronic mobility disability. Unfortunately, little is known about the feasibility and utility of pragmatic home-based exercise rehabilitation in older adults with severe mobility limitations.

The Specific Aims and Hypotheses of this proposal are:

Specific Aim #1: Using human-centered design methodologies, work with providers and patients to develop a feasible multi-component home exercise program targeting mobility, strength, and performance of task-oriented ADLs. Feasibility will be determined by assessing adherence and retention to the developed exercise program.

Hypothesis 1: The investigators hypothesize that a task-based exercise intervention can be feasibly delivered in the homes of homebound, older adults.

Specific Aim #2: Perform a feasibility study to better assess feasibility and determine the effect(s) of the home-based intervention created in Aim 1 on functional outcomes (primary outcome SPPB), mobility, and QOL changes in homebound older adults with mobility disability.

Hypothesis 2: The investigators hypothesize that the developed 12-week multi-component exercise intervention will improve performance of basic ADLs, functional mobility, and QOL; as well as outcomes related to patient satisfaction, emergency department visits, and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Veteran enrolled in the Veterans Administration Medical Health Care System's Home- Based Primary Care Program
* Aged 65 years or older

Exclusion Criteria:

* Paraplegia
* Life expectancy of less than 12 months
* Currently engaged in a physical therapy program
* Any medical condition(s) or contraindications precluding patient participation in the study as per medical judgement of study team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery | Baseline, 6 weeks, 12 weeks
  captures domains of strength, endurance, and balance and is highly predictive of disability. The SPPB score is based on timed measures of standing balance, walking speed, and ability to rise from a chair.

SECONDARY OUTCOMES:
Change in 30-second sit-to-stand test | Baseline, 6 weeks, 12-weeks
  determines lower extremity strength and endurance in older adults. The number of sit-to-stands is recorded.
Change in 30-second arm curl test | Baseline, 6 weeks, 12-weeks
  determines upper extremity strength and endurance in older adults. The number of arm curls is recorded.
Change in Grip Strength | Baseline, 6 weeks, 12 weeks
  This is a surrogate marker for sarcopenia and will be measured with a hand dynamometer. The arm to be tested held by the participant's side and elbow at a 90° angle. The participant squeezes the hand as hard as possible for few seconds. The best out of two trials separated by 60 seconds will be used.
Change in Lower Extremity Strength | Baseline, 6 weeks, 12 weeks
  will be measured with a wireless digital handheld manual muscle dynamometer during leg extension. To evaluate the knee extensor muscles, the dynamometer will be placed on the anterior part of the lower leg. Participants will perform 3 isometric maximal voluntary contractions of 5 seconds with a 60-second recovery period between contractions.

OTHER OUTCOMES:
Change in Mobility | Baseline, 6 weeks, 12 weeks
  The Activity Measure for Post-Acute Care (AM-PAC) Basic Mobility and Daily Activity Out-patient Low Functioning Short Form to assess basic mobility, daily activity, and applied cognitive.
Change in Barthel Index of Activities of Daily Living | Baseline, 6 weeks, 12 weeks
  Assesses functional dependence and independence.
Change in Life Space Activity (LAS) | Baseline, 6 weeks, 12 weeks
  A multidimensional construct that reflects the geographical area that a person moves over a period of time.
Late-Life Function and Disability Instrument (LLFDI) | Baseline, 6 weeks, 12 weeks
  Will be used to assess the subject's self-reported measures of function and disability.
Change in Quality of Life | Baseline, 6 weeks, 12 weeks
  Assessed with an analog visual scale

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Stookey, PhD, Principal Investigator — University of Maryland School of Medicine and Baltimore VA Medical Center
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers outside of our study team.